CLINICAL TRIAL: NCT04139616
Title: Prospective Validation of a Pre-Specified Algorithm for the Management of Conduction Disturbances Following Transcatheter Aortic Valve Replacement. The PROMOTE Study
Brief Title: Prospective Validation of a Pre-Specified Algorithm for the Management of Conduction Disturbances Following TAVR
Acronym: PROMOTE
Status: Recruiting | Type: Observational
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Other Study IDs: PROMOTE
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Conduction Disturbances; Transcatheter Aortic Valve Replacement; Permanent Pacemaker Implantation
Keywords: atrioventricular block; complete heart block; high-degree atrioventricular block; intraventricular conduction delay; left bundle branch block; Permanent pacemaker implantation; Right bundle branch block
MeSH Terms: conditions — Atrioventricular Block; Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- No ECG changes in patients without pre-existing RBBB: Patients with no new conduction disturbances on the ECG performed immediately post-TAVR (and no episodes of HAVB/CHB during the procedure) have a very low risk of developing HAVB/CHB or any conduction disturbance within the hours-days following the procedure. In these cases, temporary pacing will be discontinued at the end of the procedure. However, continuous ECG monitoring until hospital discharge is recommended. A 12-lead ECG is recommended 24 hours after the procedure. If no arrhythmic episodes and no ECG changes occur within the 24 hours post-procedure, the patient can be safely discharged (the day after TAVR) with no other monitoring measures in case of otherwise uneventful clinical course (absence of other TAVR related adverse events). If the patient has to remain hospitalized because of other reasons or TAVR complications, telemetry would be recommended (but no strictly required) for the detection of post-TAVR tachyarrhythmias or late ECG changes.
- Patients with pre-existing RBBB: A temporary pacing wire is recommended to be maintained for 24 hours (or at least overnight) in all patients with prior RBBB, along with telemetry and daily ECG during the entire hospitalization period (minimum of 2 days). If any ECG changes occur during the initial 2-3 days, patients can be managed according to the proposed strategy (see management strategies for groups 3 and 5). If no ECG changes or significant bradyarrythmias occur within the 2-3 days following the procedure, the patient can be discharged. Considering that the increased risk of life threatening bradyarrhythmias in these patients may extend beyond the hospitalization period, the use of continuous ECG monitoring systems (minimum of 48 hours, up to 4 weeks) may be considered.
- ECG changes in patients with prior conduction disturbances: Any significant increase in PR or QRS interval will indicate to continuing the temporary pacing for 24 hrs, with daily ECG and telemetry for 1-2 days. If the ECG changes regress in <24 hrs, an earlier removal of the temporary pacing may be considered. Also, a strategy of multiple ECGs during the first 24 hrs may be considered. If ECG changes regress or no further changes occur the patient can be discharged with no PPM at 2 days post-TAVR.
  If 24 hrs post-TAVR, the PR and QRS interval remain stable but >240 or >150 ms, respectively, and ≥20 ms longer than baseline, maintaining the temporary pacing wire for another 24 hrs is recommended. If no decrease in the PR or QRS duration occurs at day 2, the patient can be considered at risk for more advanced conduction disturbances requiring PPM. The use of an EP study may be a reasonable option for deciding PPM in those patients with prior conduction disturbances with worsening of ECG changes post-TAVR
- New-onset LBBB: Temporary pacing for 24 hrs is recommended, in all patients with new-onset LBBB post-TAVR. Earlier removal of the temporary pacing and discharged at day 1 can be considered if LBBB resolves in <24 hrs.
  If LBBB persists but no further progression of the duration of the QRS or PR interval is observed at day 1, temporary pacing can be discontinued. If no further ECG changes are observed up to day 2-3 post-TAVR, the patient can be discharged. These patients are however at increased risk of HAVB/CHB requiring PPM, and continuous ECG monitoring and/or EP studies may be considered.
  If further prolongation of the QRS or PR interval is observed at day 1, the temporary pacing is recommended for an additional 24 hrs. If the prolongation of the QRS or PR intervals continues at day 2, evaluation with EP studies or PPM implantation may be considered.
  The occurrence of any episode of HAVB/CHB following TAVR in a patient with new-onset LBBB will be considered an indication for PPM
- HAVB/CHB during the periprocedural period: Maintaining temporary pacing in patients with procedural persistent HAVB/CHB, and monitoring in intensive care unit are recommended. If HAVB/CHB persists at 24 hrs, PPM is recommended. If HAVB/CHB recovers the day after TAVR, the temporary pacing can be removed and the patient can remain hospitalized for 1 day. If another episode of HAVB/CHB occurs, PPM is recommended. If no other episode of HAVB/CHB occurs, and no other features potentially justifying PPM exist the patient can be discharged.
  Temporary pacing is recommended for 24 hrs in patients with transient HAVB during the procedure, with telemetry and daily ECG for 2 days. Discontinuing temporary pacing may be considered in those cases with brief episodes of HAVB/CHB and normal ECG. If no recurrent episodes of HAVB/CHB occur, and the patient has no other potential indications for PPM the patient can be discharged at day 2. PPM would be indicated if any recurrent episode of HAVB/CHB occurs during the hospitalization period.

SUMMARY:
The high incidence and variety of conduction disturbances post-TAVR represents a major challenge in the periprocedural management of TAVR recipients. Despite the growing body of knowledge on this topic, the large variability in the management of these complications has translated into a high degree of uncertainty regarding the most appropriate treatment of a large proportion of such patients. The implementation of a pre-specified treatment strategy translating into a more uniform practice regarding the management of conduction disturbances post-TAVR applied to a large cohort of patients would permit to identify the benefits and drawbacks of each specific aspect of the treatment algorithm proposal. This may also help to improve both the management and clinical outcomes of the complex group of patients with conduction disturbances associated with TAVR. In the end, the final objective of a pre-specified strategy for managing conduction disturbances post-TAVR should be to obtain a low rate of PPM without increasing the risk of sudden death or life threatening arrhythmic events following hospital discharge, and all this while avoiding an excessive prolongation of the hospitalization period following the TAVR procedure.

DETAILED DESCRIPTION:
The objectives of the study are:

* Feasibility: to validate and determine the applicability of a pre-specified algorithm for managing conduction disturbances in consecutive patients undergoing TAVR, also evaluating the percentage of patients included in each group of the algorithm strategy.
* Efficacy: (i) to evaluate the rate of permanent pacemaker implantation in-hospital and at 30 days compared to that of the year prior to the implementation of the protocol, (ii) to determine the incidence of sudden death at 30 days and at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

-Patients with aortic valve disease undergoing transcatheter aortic valve replacement

Exclusion Criteria:

* Prior permanent pacemaker
* Failure to provide signed informed consent for data collection
* Impossibility for a follow-up
* Unwillingness to follow the pre-specified strategy for the management of conduction disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve disease undergoing transcatheter aortic valve replacement without prior permanent pacemaker
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Rate of successful algorithm implementation and percentage of patients in each arm of the pre-specified algorithm | 1 year follow-up
Incidence of permanent pacemaker implantation | At 30-day follow-up
Incidence of permanent pacemaker implantation | At 1-year follow-up
Incidence of sudden death | At 30-day follow-up
Incidence of sudden death | At 1-year follow-up

SECONDARY OUTCOMES:
Rate, timing of and reasons for permanent pacemaker implantation | Before hospital discharge (between 1 to 30 days)
  Rate, timing of and reasons for permanent pacemaker implantation in each group of the pre-specified algorithm
Rate, timing of and reasons for permanent pacemaker implantation | At 30-day follow-up
  Rate, timing of and reasons for permanent pacemaker implantation in each group of the pre-specified algorithm
Rate, timing of and reasons for permanent pacemaker implantation | At 1 year follow-up
  Rate, timing of and reasons for permanent pacemaker implantation in each group of the pre-specified algorithm
Rate and timing of sudden death | At 30-day follow-up
  Rate and timing of sudden death in each group of the pre-specified algorithm
Rate and timing of sudden death | At 1-year follow-up
  Rate and timing of sudden death in each group of the pre-specified algorithm
Evaluation of arrhythmic events in patients with continuous ECG monitoring | After hospital discharge (up to 1-year)
  Evaluation of arrhythmic events in patients with continuous ECG monitoring at hospital discharge
Evaluation of the rate and timing of permanent pacemaker implantation | After hospital discharge (up to 1-year)
Rate of PPI among valve types | At 30-day follow-up
  Compare rate of permanent pacemaker implantation among different valve types
Rate of PPI among valve types | At 1-year follow-up
  Compare rate of permanent pacemaker implantation among different valve types
Pace dependency and pacing rate | At 30-day follow-up
  Determine the pace dependency and pacing rate in patients with periprocedural permanent pacemaker implantation (overall and in each subgroup of the algorithm)
Pace dependency and pacing rate | At 1-year follow-up
  Determine the pace dependency and pacing rate in patients with periprocedural permanent pacemaker implantation (overall and in each subgroup of the algorithm)
Factors associated with sudden death or permanent pacemaker implantation | At 30-day follow-up
  Determine factors associated with sudden death or permanent pacemaker implantation during the follow-up period overall and in each algorithm group
Factors associated with sudden death or permanent pacemaker implantation | At 1-year follow-up
  Determine factors associated with sudden death or permanent pacemaker implantation during the follow-up period overall and in each algorithm group

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puri R, Chamandi C, Rodriguez-Gabella T, Rodes-Cabau J. Future of transcatheter aortic valve implantation - evolving clinical indications. Nat Rev Cardiol. 2018 Jan;15(1):57-65. doi: 10.1038/nrcardio.2017.116. Epub 2017 Aug 24. PMID 28836620
- [Background] Kolte D, Vlahakes GJ, Palacios IF, Sakhuja R, Passeri JJ, Inglessis I, Elmariah S. Transcatheter Versus Surgical Aortic Valve Replacement in Low-Risk Patients. J Am Coll Cardiol. 2019 Sep 24;74(12):1532-1540. doi: 10.1016/j.jacc.2019.06.076. PMID 31537261
- [Background] Auffret V, Lefevre T, Van Belle E, Eltchaninoff H, Iung B, Koning R, Motreff P, Leprince P, Verhoye JP, Manigold T, Souteyrand G, Boulmier D, Joly P, Pinaud F, Himbert D, Collet JP, Rioufol G, Ghostine S, Bar O, Dibie A, Champagnac D, Leroux L, Collet F, Teiger E, Darremont O, Folliguet T, Leclercq F, Lhermusier T, Olhmann P, Huret B, Lorgis L, Drogoul L, Bertrand B, Spaulding C, Quilliet L, Cuisset T, Delomez M, Beygui F, Claudel JP, Hepp A, Jegou A, Gommeaux A, Mirode A, Christiaens L, Christophe C, Cassat C, Metz D, Mangin L, Isaaz K, Jacquemin L, Guyon P, Pouillot C, Makowski S, Bataille V, Rodes-Cabau J, Gilard M, Le Breton H; FRANCE TAVI Investigators. Temporal Trends in Transcatheter Aortic Valve Replacement in France: FRANCE 2 to FRANCE TAVI. J Am Coll Cardiol. 2017 Jul 4;70(1):42-55. doi: 10.1016/j.jacc.2017.04.053. PMID 28662806
- [Background] Auffret V, Puri R, Urena M, Chamandi C, Rodriguez-Gabella T, Philippon F, Rodes-Cabau J. Conduction Disturbances After Transcatheter Aortic Valve Replacement: Current Status and Future Perspectives. Circulation. 2017 Sep 12;136(11):1049-1069. doi: 10.1161/CIRCULATIONAHA.117.028352. PMID 28893961
- [Background] van Rosendael PJ, Delgado V, Bax JJ. Pacemaker implantation rate after transcatheter aortic valve implantation with early and new-generation devices: a systematic review. Eur Heart J. 2018 Jun 1;39(21):2003-2013. doi: 10.1093/eurheartj/ehx785. PMID 29420704
- [Background] Cerrato E, Nombela-Franco L, Nazif TM, Eltchaninoff H, Sondergaard L, Ribeiro HB, Barbanti M, Nietlispach F, De Jaegere P, Agostoni P, Trillo R, Jimenez-Quevedo P, D'Ascenzo F, Wendler O, Maluenda G, Chen M, Tamburino C, Macaya C, Leon MB, Rodes-Cabau J. Evaluation of current practices in transcatheter aortic valve implantation: The WRITTEN (WoRldwIde TAVI ExperieNce) survey. Int J Cardiol. 2017 Feb 1;228:640-647. doi: 10.1016/j.ijcard.2016.11.104. Epub 2016 Nov 9. PMID 27883975
- [Background] Rodes-Cabau J, Ellenbogen KA, Krahn AD, Latib A, Mack M, Mittal S, Muntane-Carol G, Nazif TM, Sondergaard L, Urena M, Windecker S, Philippon F. Management of Conduction Disturbances Associated With Transcatheter Aortic Valve Replacement: JACC Scientific Expert Panel. J Am Coll Cardiol. 2019 Aug 27;74(8):1086-1106. doi: 10.1016/j.jacc.2019.07.014. PMID 31439219
- [Background] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines, and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Aug 20;74(7):932-987. doi: 10.1016/j.jacc.2018.10.043. Epub 2018 Nov 6. No abstract available. PMID 30412710
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. Eur Heart J. 2012 Oct;33(19):2403-18. doi: 10.1093/eurheartj/ehs255. PMID 23026477
- [Derived] Fischer Q, Nombela-Franco L, Muntane-Carol G, Veiga G, Regueiro A, Nazif T, Serra V, Asmarats L, Ribeiro HB, Latib A, Poulin A, Cheema AN, Tirado-Conte G, Gomez-Hospital JA, Gil Ongay A, Gabani R, Arzamendi D, Brener M, Calabuig A, Scotti A, Gelain MAS, Labinaz M, Cepas-Guillen P, Cote M, Del Portillo JH, Philippon F, Rodes-Cabau J. Prophylactic Permanent Pacemaker Implantation After Transcatheter Aortic Valve Replacement. JACC Clin Electrophysiol. 2025 Nov;11(11):2484-2492. doi: 10.1016/j.jacep.2025.07.028. Epub 2025 Sep 17. PMID 40965381
- [Derived] Fischer Q, Nombela-Franco L, Muntane-Carol G, Veiga G, Regueiro A, Nazif T, Serra V, Asmarats L, Ribeiro HB, Latib A, Poulin A, Cheema AN, Jimenez-Quevedo P, Gomez-Hospital JA, Gil Ongay A, Ruberti A, Arzamendi D, Brener M, Calabuig A, Scotti A, Gelain MAS, Labinaz M, Cepas-Guillen P, Cote M, Del Portillo JH, Philippon F, Rodes-Cabau J. Risk of delayed atrioventricular block in patients without procedural conduction disturbances during transcatheter aortic valve replacement. Heart Rhythm. 2025 Apr 14:S1547-5271(25)02333-1. doi: 10.1016/j.hrthm.2025.04.017. Online ahead of print. PMID 40239910